CLINICAL TRIAL: NCT01219556
Title: Prospective, Multicentric, Large Scale Observational Study to Evaluate the Effectiveness & Safety of Xirtam H in Indian Patients Suffering From Hypertension.
Brief Title: Xirtam H Combination In the Treatment of Hypertension Evaluation Study.
Acronym: XCITE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14916; XI0911IN (Other: company internal)
Record Dates: First submitted 2010-10-07; First posted 2010-10-13 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Hypertension
Keywords: Hypertension; Antihypertensive Agents; Drug Therapy, Combination; Olmesartan Medoxomil; Hydrochlorothiazide
MeSH Terms: conditions — Hypertension | interventions — olmesartan; Hydrochlorothiazide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Olmesartan plus hydrochlorothiazide (Xirtam H, BAY98-7105)

INTERVENTIONS:
Drug: Olmesartan plus hydrochlorothiazide (Xirtam H, BAY98-7105) — Oral Xirtam H tablets every 24 hours (Q24H) or as per prescribing information

SUMMARY:
This is post-marketing observational study in which data on safety and effectiveness of Xirtam H will be collected from routine clinical practice. The study objectives are to investigate the effect of Xirtam-H on blood pressure and achievement of target blood pressure as well as safety and satisfaction of treatment. All hypertensive patients (Blood pressure > 140/90 mmHg) where investigator feels that addition of Xirtam H would be beneficial to patients will be included in non interventional study. The routine investigation suggested by the attending physician will be done in patients of hypertension. No additional investigation will be done for the study purpose. The patient not controlled on existing treatment and prescribed Xirtam H will be included in study after taking the informed consent. The patient will be followed up for 2-follow up visit each after 6 weeks. The physical examination, routine investigation, blood pressure measures will be done and the data will be entered in the CRF as mentioned in CRF in each visit. The study is planned to be carried out in 9604 patients from around 300 - 350 trial sites in India.

ELIGIBILITY:
Inclusion Criteria:

* All Indian hypertensive patients (Blood pressure > 140/90 mm Hg) where investigator feels that addition of Xirtam H would be beneficial to patients will be included in non interventional study.

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with corresponding product prescribing information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertension
Sampling Method: Probability Sample
Enrollment: 8704 (Actual)
Dates: Start 2010-11; Primary Completion 2012-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Changes in seated diastolic pressure | 12 weeks
Changes in seated systolic pressure | 12 weeks
Achievement of target blood pressure as per Sixth Report of the Joint National Committee of High Blood Pressure (JNC-VII) | 12 weeks

SECONDARY OUTCOMES:
Number of patients with adverse events as measure of safety | 12 weeks
Percentage of patients with satisfaction to treatment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, India